CLINICAL TRIAL: NCT06035653
Title: A Step Towards Fully Automated Adaptive Radiotherapy in Head & Neck Cancer: A Human Versus Machine Comparison Study
Brief Title: A Human Versus Machine Comparison Study
Acronym: HuVeM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: East and North Hertfordshire NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: RD2021-57
Record Dates: First submitted 2023-05-09; First posted 2023-09-13 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A: Minimum of 12 patients who required total radiotherapy replan
- B: Minimum of 28 patients who were reviewed in the multi-professional meeting but did not require full replan

SUMMARY:
The study aims to retrospectively, and anonymously analyse the data of patients treated over a period of 12 months. These are the patients whose radiotherapy plan were needed to be reviewed in the weekly on-treatment head and neck multi-professional radiotherapy meeting during the course of their radiation.

Collected clinical data will be included in the retrospective analysis, comparing the clinical decision (gold standard of care), against the predictive capability of intelligence software

DETAILED DESCRIPTION:
This is a single centre, non-interventional study comparing "machine" against clinician's standard of care approach. The utilisation of intelligence software is for research purposes only and does not permit active changes to patients' clinical management. Any software related analyses will be done after patients have completed radiation treatment.

All consented patients who were discussed in the head and neck CBCT meeting and deemed to require new masks / recontouring / replanning - Cohort A will be analysed on completion of radiotherapy. These patients typically are ones with nodal disease of >3cm at presentation, and whose weight change is notable 5 - 10% of baseline in the first 2 weeks of their treatment. There have been 28 patients in 12 months previously.

Other patients discussed in the head and neck CBCT meeting on completion of radiation - Cohort B, whose radiotherapy was not deemed to require total replan but were clinically deemed 'marginal' will be included. These patients tend to be ones with weight loss measuring close to 1.29cm lateral separation or between the skin surface and the head shell.

The radiotherapy replan volumes CTVs of Cohort A patients will retrospectively compared to the CTVs produced by the intelligence software. The time using the software to produce dynamic CTVs will be compared with the time needed for the clinicians to create new CTV for the radiotherapy replan, which will be recorded prospectively.

The CBCTs of both Cohorts A & B will be analysed using the intelligence software to determine the adequacy of PTV coverage. This is to be compared with the departmental quality assurance/audit of PTV margins.

The software will also be used to calculate various aspects of the radiotherapy plans, including the cumulative dose distribution over the period of dynamic anatomical change Cohorts A & B.

ELIGIBILITY:
Inclusion Criteria:

* i. Head and neck cancer patients who require new mask for radiotherapy replanning will be included (Cohort A). These patients typically are ones with rapid shrinkage of the nodal disease, or whose weight change is notable (5 - 10% of baseline) in the first 2 weeks of radiotherapy ii. Patients on close observation of the head and neck multi-professional team but whose radiotherapy did no undergo total replan treatment will be included (Cohort B)

Exclusion Criteria:

i. Patients whose primary malignancy is not of head and neck origin ii. Patients who specifically opt against their information be used anonymously iii. Head and neck cancer patients whose radiotherapy plans did not require review in the head and neck multi-professional radiotherapy meeting iv. Patients under the age of 18

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Minimum of 12 patients who required total radiotherapy replan (Cohort A) Minimum of 28 patients who were reviewed in the multi-professional meeting but did not require full replan (Cohort B) Minimum of 40 patients in total (Cohorts A&B).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2023-11-27 (Estimated); Study Completion 2023-11-27 (Estimated)

PRIMARY OUTCOMES:
Interobserver variability studies (IOV) between manually contoured CTVs and software-generated deformed CTVs | 1 year
  Measured by volume differences
Interobserver variability studies (IOV) between manually contoured CTVs and software-generated deformed CTVs - Sorensen-DICE Coefficient | 1 year
  Measurement of ratio of overlap
Interobserver variability studies (IOV) between manually contoured CTVs and software-generated deformed CTVs - Discordance Index | 1 year
  Measurement of over contouring
Interobserver variability studies (IOV) between manually contoured CTVs and software-generated deformed CTVs - Geographical miss index | 1 year
  Measurement of under contouring
Interobserver variability studies (IOV) between manually contoured CTVs and software-generated deformed CTVs - Hausdorff distance | 1 year
  Measurement of distance between 2 volumes
PTV margins compared against the departmental standards | 1 year
  Proportion of clinical tumour volume covered by different radiotherapy set up margins 3, 4 and 5mm

SECONDARY OUTCOMES:
Potential time saved recontouring with software and the associated cost of re-planning adaptive radiotherapy | 1 year
  Difference between time spent on re- contouring and time spent on editing software deformed CTVs
Evaluation of clinical decision on total radiotherapy re-plan | 1 year
  Measured by retrospective assessment of dose accumulation of the CTVs

CONTACTS AND LOCATIONS:
Locations (1):
- East & North Hertfordshire NHS Trust, Northwood, UK, United Kingdom

IPD SHARING:
Plan to Share IPD: No